CLINICAL TRIAL: NCT01750684
Title: A Phase 2 Double-blind, Randomized, Placebo-controlled Study to Determine the Safety, Tolerability and Potential Activity of AC105 Following a Regimen of 6 Doses Over 30 Hours in Patients With Acute Traumatic Spinal Cord Injury (SCI).
Brief Title: AC105 in Patients With Acute Traumatic Spinal Cord Injury
Acronym: AC105
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated by the Sponsor due to insufficient enrollment.
Sponsor: Acorda Therapeutics (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); DP Clinical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACPM-SI-1009
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Acute Spinal Cord Injury
Keywords: Acute; Traumatic; SCI; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): Patients randomized (1:1) to the placebo arm will receive an initial intravenous infusion of saline for 30 minutes within a pre-specified time window (12, 9, 6 hours post-injury). Patients will receive 5 additional infusions of the same dose and duration at 6 -hour intervals.
  Interventions: Other: Placebo
- AC105 (Active Comparator): Patients randomized (1:1) to the active drug arm will receive an initial intravenous infusion of AC105 for 30 minutes within a pre-specified time window (12, 9, 6 hours post-injury). Patients will receive 5 additional infusions of the same dose and duration at 6 -hour intervals.
  Interventions: Drug: AC105

INTERVENTIONS:
Drug: AC105
  Arms: AC105
Other: Placebo
  Arms: Saline

SUMMARY:
The principal aim of this study was to establish the feasibility of rapid administration, safety, and tolerability of AC105 in patients with acute spinal cord injury.

DETAILED DESCRIPTION:
To determine safety and tolerability of AC105 following a regimen of 6 intravenous doses over 30 hours in patients with acute non-penetrating traumatic spinal cord injury (SCI).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age, inclusive
* Acute traumatic SCI, at a neurological level between C4 and T11
* No evidence of penetrating or transection injury (e.g. caused by projectile or stab wound)
* Neurological ASIA Impairment Scale A, B or C
* Patient is able to provide written or verbal witnessed consent. If unable to provide either, consent may be provided by legally authorized representative (LAR)
* Patient is able to initiate treatment within time window of injury

Exclusion Criteria:

* Known allergy or hypersensitivity to polyethylene glycol
* Mental impairment or other conditions that would preclude a reliable ASIA exam or adequate consent
* Positive urine pregnancy test result
* Serum creatinine level ≥ 2 mg/dL
* History or active renal failure or dialysis
* Mean arterial blood pressure < 60 mmHg despite vasopressor treatment
* On a current regimen of digoxin
* Chronic use of magnesium salts prior to the SCI (within 1week of presentation) and/or the use of magnesium salts in the acute care setting prior to the administration of investigational product
* Any other medical condition that, in the judgment of the investigator, would preclude provision of informed consent, make participation in the study unsafe, or unreasonably complicate follow-up or the interpretation of study outcome data or may otherwise interfere with achieving the study objectives
* In the judgment of the Investigator, cannot adequately provide informed consent, is likely to be non-compliant, or may be unable to cooperate with study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Eisen, MD, Study Director — Acorda Therapeutics

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 subjects were enrolled. 2 subjects randomized to placebo were subsequently deemed ineligible and were not treated with the investigational product; they were excluded from the analysis. A total of 13 subjects received at least 1 infusion of the investigational product (AC105 and placebo) and were included in the Safety Population.
Groups:
- Placebo: Patients randomized (1:1) to the placebo arm will receive an initial intravenous infusion of saline for 30 minutes within a pre-specified time window (12, 9, 6 hours post-injury). Patients will receive 5 additional infusions of the same dose and duration at 6 -hour intervals.
  Placebo
- AC105: Patients randomized (1:1) to the active drug arm will receive an initial intravenous infusion of AC105 for 30 minutes within a pre-specified time window (12, 9, 6 hours post-injury). Patients will receive 5 additional infusions of the same dose and duration at 6 -hour intervals.
  AC105
Period: Overall Study
Arm/Group | Placebo | AC105
Started | 6 | 7
Completed | 4 | 5
Not Completed | 2 | 2
Not completed — Death | 1 | 0
Not completed — Non-compliance with Study Drug | 0 | 1
Not completed — Withdrawn by Sponsor | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AC105 | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (7.12) | 38.3 (6.23) | 37.7 (4.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Treatment-Emergent Adverse Events (TEAEs) are defined as AEs with date time of onset (or worsening) on or after the start date time of the first infusion and no more than 30 days after the end of the last infusion.
Time Frame: up to 6 months
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | AC105
Number analyzed (Participants) | 6 | 7
participants
  Mild TEAEs | 4 | 6
  Moderate TEAEs | 3 | 5
  Severe TEAEs | 2 | 3
  Serious TEAEs | 1 | 2
  Drug-related TEAEs | 0 | 2
  TEAEs Leading to Death | 1 | 0

2. Secondary Outcome: Pharmacokinetic (PK) Parameters of AC105 Using Individual Patient Plasma Concentration-time Data
Description: Measuring Maximum Measured Plasma Concentration (Cmax), Time to Maximum Measured Plasma Concentration (Tmax), Half-life calculated as In(2)/kel (T 1/2) and Area Under the Plasma Concentration versus time curve (AUC).
Time Frame: baseline, prior to and up to 5 hours following last infusion
Population: No subjects were analyzed. No data was collected. There was a change in the planned analysis to not perform formal PK analysis for a terminated study and abbreviated Clinical Study Report.
Groups:
- Saline: Patients randomized (1:1) to the placebo arm will receive an initial intravenous infusion of saline for 30 minutes within a pre-specified time window (12, 9, 6 hours post-injury). Patients will receive 5 additional infusions of the same dose and duration at 6 -hour intervals.
  Placebo
Arm/Group | Saline | AC105
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months.
Description: TEAEs are defined as adverse events (AEs) with date time of onset (or worsening) on or after the start date time of the first infusion and no more than 30 days after the end of the last infusion. Adverse events were classified according to Version 16.0 of the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary.
Arm/Group | Placebo | AC105
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/7
Other Adverse Events (participants affected / at risk) | 4/6 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | AC105 (N=7)
Pneumonia (Infections and infestations) | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | AC105 (N=7)
Nausea (Gastrointestinal disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 2 | 3
Pneumonia (Infections and infestations) | 2 | 3
Depression (Psychiatric disorders) | 3 | 2
Hypotension (Vascular disorders) | 2 | 2
Neuralgia (Nervous system disorders) | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Ileus (Gastrointestinal disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 2
Oxygen saturation decreased (Investigations) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Neurogenic bowel (Gastrointestinal disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.